CLINICAL TRIAL: NCT00332761
Title: An 8-Week Randomized, Double-Blind, Placebo-Controlled Trial Examining The Efficacy And Safety Of Caduet® In Simultaneously Achieving Blood Pressure And Lipid Goals In An Untreated Hypertensive And Dyslipidemic Subject Population. (CUSP - Caduet in Untreated Subject Population)
Brief Title: Caduet in an Untreated Subject Population
Acronym: CUSP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3841046
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Hypertension; Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — amlodipine, atorvastatin drug combination

INTERVENTIONS:
Drug: Caduet

SUMMARY:
The purpose of this study is to determine if Caduet will lower blood pressure to <140/90 mmHg and lower LDL Cholesterol to <100 mg/dL in subjects with hypertension and dyslipidemia who are not currently being treated for these medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were recently diagnosed with both hypertension and dyslipidemia and who are not yet taking any medications for these conditions OR subjects with both hypertension and dyslipidemia who were previously treated with antihypertensive and/or lipid lowering medications but discontinued these medications for at least 3 months prior to the Screening visit.
* SBP 140-169 mmHg and/or DBP 90-105 mmHg, LDL-C 110-160 mg/dL

Exclusion Criteria:

* Subjects with a history of MI, angina, coronary artery bypass or intra-coronary interventions, stroke, TIA, CHF or cardiomyopathy requiring treatment.
* Subjects with a known history of Type I or Type 2 Diabetes Mellitus or a fasting blood glucose > 126 mg/dL at the Screening visit.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2006-06; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects achieving both blood pressure goal (<140/90 mmHg) and LDL-C goal (<100 mg/dL) at Week 4.

SECONDARY OUTCOMES:
The percentage of subjects achieving both blood pressure goal (<140/90 mmHg) and LDL-C goal (<100 mg/dL) at Week 8.
Change from Baseline to Week 4 in SBP, DBP, and Framingham 10-year CHD risk score.
Percent change from Baseline to Week 4 in LDL-C, HDL, TC, and TG.
The percentage of study subjects achieving each of the following goals at Week 4: SBP, DBP, and LDL-C.
Change from Baseline to Week 8 in SBP, DBP, and Framingham 10-year CHD risk score.
Percent change from Baseline to Week 8 in LDL-C, HDL, TC, and TG.
The percentage of study subjects achieving each of SBP, DBP, and LDL-C goals at Week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- United States (33):
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Garden Grove, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Aventura, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Bossier City, Louisiana
  - Pfizer Investigational Site, Fair Haven, Michigan
  - Pfizer Investigational Site, Livonia, Michigan
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Excelsior Springs, Missouri
  - Pfizer Investigational Site, Berlin, New Jersey
  - Pfizer Investigational Site, Elizabeth, New Jersey
  - Pfizer Investigational Site, Princeton, New Jersey
  - Pfizer Investigational Site, South Bound Brook, New Jersey
  - Pfizer Investigational Site, Binghamton, New York
  - Pfizer Investigational Site, Monroe, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Bensalem, Pennsylvania
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Colleyville, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Temple, Texas
  - Pfizer Investigational Site, Norfolk, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3841046&StudyName=Caduet%20in%20an%20Untreated%20Subject%20Population.